CLINICAL TRIAL: NCT05062603
Title: Prospective Observational Study Looking at Lung Ultrasound Changes During Recovery From COVID19 Infection
Brief Title: Lung Ultrasound Changes in Covid 19 Patients Discharged From Hospital
Status: Completed | Type: Observational
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: C&W20/036; IRAS number 286015 (Other: Integrated Research Application System)
Record Dates: First submitted 2021-09-29; First posted 2021-09-30 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Covid19; Coronavirus; Coronavirus Infection; SARS-CoV Infection
Keywords: Coronavirus; COVID-19; Lung ultrasound; Respiratory
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lung ultrasound has been used to help diagnose COVID-19 as an alternative to CT scanning and chest X-ray. CT scanning is onerous and there are difficulties taking critically unwell patients there as well as decontamination issues.

Chest X-ray misses up to 40% of COVID diagnoses. Although lung ultrasound can diagnose, the investigators do not know how long these lung ultrasound changes last. The investigators would like to follow up patients to characterise the pattern of changes and how long they last. This is particularly important given a potential second surge of COVID-19 is looming and the investigators would like to know if lung ultrasound changes are new or old in patients presenting during this second wave and in the future.

DETAILED DESCRIPTION:
Ultrasound has been invaluable during this pandemic to diagnose COVID-19. The investigators have used it alongside CT scanning to rationalise the number of CT scans especially when patients are unstable. The investigators do not know how long these changes last on lung ultrasound after discharge and the investigators wish to study this.

This is because patients will start presenting shortly who have a history of COVID-19 with acute medical problems and if the investigators are to use lung ultrasound again the investigators would like to know whether the changes the investigators see are new or old.

This is vitally important before a second surge and especially so before winter. This may also facilitate triage of patients from the front door in the Emergency department to different areas (such as COVID-19 zones or clean areas).

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Confirmed COVID-19 positive with changes on CXR or CT scan
* Having had an initial lung ultrasound in the Emergency department when they were first admitted into the hospital.

Exclusion Criteria:

* Pre-existing lung disease
* Heart failure
* Under 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with a confirmed COVID-19 viral infection.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Assessment of lung ultrasound changes over the time period of follow up. | Approximately 3 months or until the ultrasound changes in the lung had normalised
  The assessment will determine how long it takes for lung ultrasound changes to resolve following discharge from hospital in patients who were diagnosed with COVID-19 (unit of measurement: days).

SECONDARY OUTCOMES:
Exploration of ongoing symptoms | Approximately 3 months or until the ultrasound changes in the lung had normalised
  Ongoing symptoms will be explored by using screening questions.

CONTACTS AND LOCATIONS:
Overall Officials: Paramjeet Deol, MBChB FRCEM, Principal Investigator — Chelsea and Westminster NHS Foundation Trust
Locations (1):
- Chelsea and Westminster Hospital, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Poggiali E, Dacrema A, Bastoni D, Tinelli V, Demichele E, Mateo Ramos P, Marciano T, Silva M, Vercelli A, Magnacavallo A. Can Lung US Help Critical Care Clinicians in the Early Diagnosis of Novel Coronavirus (COVID-19) Pneumonia? Radiology. 2020 Jun;295(3):E6. doi: 10.1148/radiol.2020200847. Epub 2020 Mar 13. No abstract available. PMID 32167853
- [Background] Huang Yi, Sihan Wangm Yue Liu, Yaohui Zhang, Chuyun Zheng, Yu Zheng, CHaoyang Zhangm et al. A preliminary study on the ultrasonic manifestations of Peripulmonary lesions of non-critical Novel Coronavirus Pneumonia (Covid-19).
- [Background] Peng QY, Wang XT, Zhang LN; Chinese Critical Care Ultrasound Study Group (CCUSG). Findings of lung ultrasonography of novel corona virus pneumonia during the 2019-2020 epidemic. Intensive Care Med. 2020 May;46(5):849-850. doi: 10.1007/s00134-020-05996-6. Epub 2020 Mar 12. No abstract available. PMID 32166346